CLINICAL TRIAL: NCT06011590
Title: QRS Microfragmentation in ECG as Predictor of Mortality and Morbidity - a Retrospective Analysis
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 1244/2022
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Risk Stratification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: All patients treated at the Department of Internal Medicine at the Medical University of Innsbruck between 01.01.2000 and 31.07.2022, in whom a 10 second 12-lead ECG is available from clinical routine.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — No intervention.

SUMMARY:
Over the past decades, several ECG-based parameters have been identified as independent predictors of worsened prognosis in affected patients. In addition to visual assessment of morphology, methods of computer-based machine ECG analysis have gained importance in recent years. These methods allow the detection of systemic abnormalities in ECGs that are not visible to the naked eye. An example of this is provided by the so-called "QRS microfragmentations".

The aim of this evaluation is to retrospectively collect all established as well as new quantitative and qualitative ECG parameters (such as QRS microfragmentation) in a large patient collective. Subsequently, after characterization of the patients, an independent multivariate risk prediction model should be developed based on computer-based ECG analysis using maschnine learning algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented to the Department of Internal Medicine at the Medical University in Innsbruck between 01.01.2000 and 31.07.2022 and received an ECG recording as part of routine clinical practice.
* Age ≥ 18 years
* Residence in Austria

Exclusion Criteria:

* Insuffizient ECG Recording quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who presented to the Department of Internal Medicine at the Medical University in Innsbruck between 01.01.2000 and 31.07.2022 and received an ECG recording as part of routine clinical practice.
Sampling Method: Probability Sample
Enrollment: 150000 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
All cause mortality | between 01.01.2000 and 31.07.2022
  Death of any cause

SECONDARY OUTCOMES:
Hospitalization | between 01.01.2000 and 31.07.2022
  Unplanned Hospitalization
Lenght of hospital stay | between 01.01.2000 and 31.07.2022
  Lenght of hospital stay

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon reasonable request and after concluding all legal and ethic formalities.